CLINICAL TRIAL: NCT05565443
Title: A Phase I/II Study for Bilateral Putamenal Delivery of Recombinant Glucocerebrosidase in Patients With Parkinson's Disease Using MR-guided Focused Ultrasound Induced Opening of the Blood-brain Barrier
Brief Title: MR-guided Focused Ultrasound Plus GCase
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PD016
Record Dates: First submitted 2022-09-07; First posted 2022-10-04 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Parkinsons Disease
Keywords: Parkinson's disease; Glucocerebrosidase; GCase
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A two-arm, open-label, intervention only clinical study. One arm to enroll 7 GBA PD patients, the second arm to enroll 7 idiopathic PD patients. The study involves focused ultrasound procedures targeting bilateral putamen in patients with Parkinson's Disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Idiopathic PD Patients (Experimental): Idiopathic PD patients receiving 3 cycles of BBBO. There is option to include simultaneous GCase delivery after safety profile review by Data and Safety Monitoring Board (DSMB).
  Interventions: Device: Blood Brain Barrier Disruption - Functional
- GBA PD Patients (Experimental): GBA PD patients receiving 3 cycles of BBBO. There is option to include simultaneous GCase delivery after safety profile review by Data and Safety Monitoring Board (DSMB).
  Interventions: Device: Blood Brain Barrier Disruption - Functional

INTERVENTIONS:
Device: Blood Brain Barrier Disruption - Functional — Delivery of GCase across the BBB to form a disease modifying strategy for patients with Parkinson's Disease

SUMMARY:
The goal of this study is to establish safety and feasibility of intracerebral delivery of GCase via MRgFUS. This technique may offer potential benefits given the exposure of the putamen to GCase in animal models has been shown to be efficacious in improving Parkinson's disease pathology and phenotype.

DETAILED DESCRIPTION:
This is a two-arm, open-label, intervention only phase I/II clinical study. One arm of the study will enroll seven (7) GBA PD patients and the other arm seven (7) idiopathic PD patients. During the intervention phase, the first four subjects of each arm will receive three transcranial bilateral putamenal GCase at 30 IU/kg IV every two weeks, followed by 60 IU/kg in the next three subjects. Following three treatments in this study, the subjects will be followed for twelve months.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between age 35 and 80 years, inclusive.
* Able and willing to give informed consent.
* Diagnosis of PD satisfying MDS Clinical Diagnostic Criteria for PD
* At least 2 years from initial diagnosis
* Hoehn and Yahr Stage 1-3 on PD medication
* Dopaminergic deficit by a positive DAT SPECT scan
* On stable regimen of PD medications for at least 90 days prior to the study
* American Society of Anesthesiologists (ASA) score 1-3
* Harbor at least one GBA mutation if enrolled in the GBA PD arm or two wild-type GBA alleles if enrolled in the idiopathic PD arm

Exclusion Criteria:

* Positive pregnancy test (for pre-menopausal women).
* Contraindication to DEFINITY ultrasound contrast agent or perflutren (e.g. hypersensitivity, known left or bidirectional cardiac shunt)
* Contraindication to MRI or gadolinium-DTPA (e.g. incompatible device, hypersensitivity)
* Insulin-dependent diabetes mellitus that is not well-controlled or that in the Investigator's opinion precludes participation in the study.
* Severely impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2 and/or on dialysis.
* Currently participating in another clinical therapeutic trial
* Patient receiving bevacizumab (Avastin) therapy
* Subjects with evidence of cranial or systemic infection.
* Cerebral or systemic vasculopathy.
* Documented cerebral infarction within the past 12 months or TIA in the past 1 month.
* Contraindication to GCase enzyme therapy, specifically previous hypersensitivity reaction to GCase enzyme therapy
* Parkinsonism plus symptoms, secondary parkinsonism
* Previous neurosurgical procedure for PD

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 12 Months
  Measure of the adverse events through the intervention phase and follow-up. All adverse events and/or Serious Adverse Events will be documented and reported according to CTCAE criteria.

SECONDARY OUTCOMES:
Feasibility of MRgFUS BBB opening for GCase brain delivery | 12 Months
  Using MRI images to measure:
  1. The qualitative measure of the MRI T1-weighted with gadolinium of contract extravasation in the sonicate putamen.
  2. The qualitative measure of the dynamic contrast enhanced (DCE) MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Sunybrook Research Institute, Toronto, Ontario, Canada